CLINICAL TRIAL: NCT04689633
Title: Ultrasound-guided Bilateral Quadratus Lumborum Block Versus Erector Spinae Block for Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: Quadratus Lumborum Block Versus Erector Spinae Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shadwa Rabea Mohamed, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 135-12/2018
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus lumborum block (Active Comparator): received bilateral ultrasound-guided Quadratus lumborum block using 20 ml bupivacaine 0.25% on each side
  Interventions: Procedure: nerve block
- Erector spinae block (Active Comparator): received bilateral ultrasound-guided erector spinae block using 20 ml bupivacaine 0.25% on each side
  Interventions: Procedure: nerve block
- Control (No Intervention): didn't received any block

INTERVENTIONS:
Procedure: nerve block — bilateral ultrasound-guided posterior quadratus lumborum block was done in the lateral decubitus and linear or curvilinear probe was used according to the depth and placed in the midaxillary line in the transverse plane above the iliac crest
  Arms: Erector spinae block; Quadratus lumborum block

SUMMARY:
The patients were randomly allocated into 3 parallel groups of 20 patients in each group by using computer generated tables. group(Q):received bilateral sonar-guided quadratus lumborum bolck using 20 ml bupivacaine 0.25%on each side.group(E): received bilateral ultrasound-guided erector spinae block using 20 ml bupivaciane 0.25%on each side. group(C):didn't received any block

DETAILED DESCRIPTION:
on arrival to the operative room all patients were monitored with standared monitoring. then IV cannula were inserted. preoxygenation with 100% oxygen and induction of GA by 1mic/kg fentanyl and 2 mg/kg of 1%propofol. endotracheal intubation was facilitated by 0.5mg/kg of atracurium. isoflurane 1-2% with oxygen was used for anesthetic maintenance and 0.15 mg/kg intermittent doses of atracurium to maintain adequate muscle relaxation. ventilation was controlled to maintain end tidal CO2 at 35-40 mmHg and SaO2 between 95-100. after stabilization of the patient's hemodynamics and before surgical incision, quadratus lumborum and erector Spinae block were performed according to patient's group by the same anesthetist with the patient in lateral or prone position respectively.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists(ASA) physical status1and2 scheduled for elective cholecystectomy under general anesthesia

Exclusion Criteria:

* Allergy to studed drugs
* morbid obesity
* patient refusal
* infection at the side of the bolck
* emergency laparoscopic cholecystectomy
* if laparoscopic procedure converted to open

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
time of first postoperative analgesic request | 24 hours
  first time that patient need analgesia and visual analogue scale more than 3

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Hassaneen, MD, Study Chair — Assistant professor
Locations (1):
- Faculty of Medicine, Minya, Egypt